CLINICAL TRIAL: NCT00459576
Title: Risk of Asthma in Infants With Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Indiana University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Other Study IDs: 0211-15
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Asthma; Eczema; Dermatitis, Atopic
Keywords: Asthma; Eczema; Dermatitis, Atopic; Infant
MeSH Terms: conditions — Asthma; Eczema; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We have retained nasal cell samples, whole blood cells, and serum.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Infants will be enrolled in this study if they have never been diagnosed with asthma or wheezing and have been diagnosed with atopic dermatitis or eczema. Infants with some types of skin rashes are at high risk for developing asthma by 6 years of age. The purpose of this study is to determine whether we can identify infants who will develop asthma.

DETAILED DESCRIPTION:
Asthma is a disease characterized by recurrent episodes of wheezing, inflammation of the airways, and airways that are very sensitive to stimulation (hyper-responsiveness). Symptoms of asthma frequently begin in early childhood; however, it has been difficult to identify pre-symptomatic, at-risk infants and toddlers. Family history of asthma and allergy is strongly associated with the early onset and persistence of asthma symptoms, and children with early onset persistent asthma are more likely to demonstrate allergies. The development of allergic disease results from complex interactions between genetic susceptibility and environmental factors; however, infants with atopic dermatitis have a 50% chance of developing asthma by 6 years of age. Airway inflammation and airway hyper-responsiveness are characteristics of asthmatic children. We plan to evaluate whether infants with allergic dermatitis have evidence of airway inflammation and hyper-responsiveness, and whether cells from the blood and the nose are also hyper-responsive to stimulation prior to the onset of clinical symptoms of asthma. In addition we will evaluate whether certain genetic profiles are associated with allergic disease in infants.

ELIGIBILITY:
Inclusion criteria-

1. Full term infants born greater than 37 weeks
2. History of atopic dermatitis or eczema

Exclusion criteria

1. Heart disease
2. asthma
3. Respiratory illness such as RSV, bronchiolitis or croup
4. Hospitalization for respiratory illness
5. History of wheezing

Ages: 2 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Our population was recruited through primary physician, pediatric practices, and dermatology groups through out Indianapolis Indiana and the surrounding counties. We also ran ads in local newspapers.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2005-05; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Tepper, MD, PhD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States